CLINICAL TRIAL: NCT06772090
Title: A Randomized Placebo-controlled Feasibility Trial of Probiotic Supplementation During Adjuvant or Neoadjuvant Cytotoxic Chemotherapy for Solid Tumor Malignancies
Brief Title: Probiotic Supplementation During Cytotoxic Chemotherapy for Solid Tumor Malignancies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023LS220
Record Dates: First submitted 2025-01-02; First posted 2025-01-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumor, Adult; Cytotoxicity
MeSH Terms: interventions — Lacteol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 0: Placebo (Placebo Comparator): The placebo will also be manufactured and provided by the commercial provider.
  Interventions: Other: Placebo
- Phase 1: Placebo (Placebo Comparator): Placebo capsules of the same size and shape to be taken daily for 12 weeks. The placebo will also be manufactured and provided by the commercial provider.
  Interventions: Other: Placebo
- Phase 1: Treatment (Active Comparator): 50 billion CFU of a commercially available Lactobacillus and Bifidobacterium oral capsule, to be taken daily for 12 weeks
  Interventions: Biological: Lactobacillus and Bifidobacterium

INTERVENTIONS:
Biological: Lactobacillus and Bifidobacterium — Each lot of Lactobacillus and Bifidobacterium and placebo capsules to be used in this study will undergo bioburden testing (tested as per USP <61>) to ensure that each lot has:
  * Not more than 2000 colony forming unit (CFU) of contaminating (other than the seven strains of bacteria used in the Lactobacillus and Bifidobacterium capsules) aerobic bacteria per gram or dose (whichever is greater);
  * Not more than 200 CFU of yeasts and molds per gram or dose (whichever is greater); and
  * No bile-tolerant Gram-negative bacteria, Escherichia coli, Salmonella species (in 10 gm), Pseudomonas aeruginosa, Staphylococcus aureus, and Clostridium species per gram or dose (whichever is greater; tested as per USP<62>).
  Arms: Phase 1: Treatment
Other: Placebo — Placebo capsule manufactured in same facility as experimental capsule.
  Arms: Phase 0: Placebo; Phase 1: Placebo

SUMMARY:
This is a pilot single-blind placebo-controlled randomized trial to establish experimental feasibility. We plan on enrolling a pilot cohort of 40 patients, with up to 5 patients in treatment phase 0 and the remaining in treatment phase I. During Phase I, the remaining participants will be assigned to either treatment or control group using dynamic block randomization balancing on sex, age group, and disease histology.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old
* Diagnosis of stage III colon cancer
* Undergoing chemotherapeutic treatment within the MHFV or MVAHC medical systems.

Exclusion Criteria:

* Allergy or sensitivity to probiotic supplementation
* Diagnosis/history of:

Non-colon GI cancer or chronic GI-related disease or disorders such as gastric ulcer, irritable bowel syndrome, inflammatory bowel disease, or intestinal malabsorption syndrome Cognitive impairment, such as dementia, or developmental disorder that would affect ability to give consent or comply with study procedures

* Current treatment of cancer other than non-melanoma skin cancer, including metastases and recurrences
* Current participation in another interventional study of medication(s)
* Major changes in eating habits within the past 3 months, such as stopping or starting a restricted diet
* BMI ≥40 kg/m2 or ≤17 kg/m2
* Unexpected change in weight of ˃4.5 kg within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-12-25 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants at end of study | Week 12
  Determine the feasibility of conducting a randomized, placebo controlled clinical trial of probiotic supplementation in patients with solid tumor malignancies undergoing cytotoxic chemotherapeutic treatment. Number of participants that completed the study.

SECONDARY OUTCOMES:
Number of Adverse Events related to Cytotoxic Chemotherapy | Week 12
  To evaluate how probiotic supplementation impacts cytotoxic chemotherapy-associated GI toxicities, including nausea, anorexia, and diarrhea. Number of adverse events correlated to nausea, anorexia or diarrhea.